CLINICAL TRIAL: NCT01539967
Title: Is the Residual Gastric Volume After Sleeve Gastrectomy an Objective Criterion to Adapt the Treatment Strategy After Failure?
Brief Title: Impact of the Residual Gastric Volume in Laparoscopic Sleeve Gastrectomy's Failure
Acronym: GASTROMANCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI09-PR-REGIMBEAU; 2009-A00603-54 (Other: ID-RCB)
Record Dates: First submitted 2012-02-07; First posted 2012-02-28 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Laparoscopic Sleeve Gastrectomy; Obesity follow-up
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Laparoscopic Sleeve Gastrectomy — the operative technique consists in few steps:
  * position of 4 trocars and insertion of a nasogastric tube
  * dissection and mobilization of the greater curvature of the stomach
  * preparation of the stomach for division
  * gastric partition
  * extraction of the gastric remnant
  * postoperative surveillance

SUMMARY:
Obesity is a worldwide health problematic whose incidence is increasing especially in developed countries. The surgical management of this illness consists in different techniques such as Laparoscopic Sleeve Gastrectomy but this treatment could not be efficient enough. The causes of failure after Laparoscopic Sleeve Gastrectomy are not known but could include the residual gastric volume.

The aim of the present study was to determine whether the residual gastric volume is involved in Laparoscopic Sleeve Gastrectomy's failure.

DETAILED DESCRIPTION:
This study can be done in three steps:

1. From a prospective database, patients are selected if they were operated by Laparoscopic Sleeve gastrectomy at least two years before.
2. these patients are convoked by their surgeon, who proposed them to participate at this study. During this consultation, the BAROS score is calculated by the surgeon and reported in the case report form of the patient.
3. After checking the possible contraindication, a gastric computed tomography volumetry is done and the residual gastric volume is calculated by two independent radiologists.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* laparoscopic Sleeve gastrectomy performed two years before
* surgery performed in the digestive surgery department of the Amiens University Hospital

Exclusion Criteria:

* pregnancy or breastfeeding
* death of the patient or lost of follow-up
* patient under legal or administrative protection
* contraindication to the volumetry (pregnancy, technical impossibility)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
calculation of the BAROS Score | during the consultation two years after the surgery
  the BAROS Score is calculated by the surgeon and corresponds to the presence of a failure of Laparoscopic Sleeve Gastrectomy

SECONDARY OUTCOMES:
measure of the residual gastric volume by the radiologists | two years after the surgical procedure
  the residual gastric volume is measured by gastric computed-tomography volumetry two years after Laparoscopic Sleeve Gastrectomy and is defined as the volume held between the gastro-oesophageal junction and the pylorus. Two radiologists interpreted the volumetry and conflicts between the 2 observers are resolved by consensus: the larger of each patient's two volume determinations was considered as being closest to the true residual gastric volume

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc REGIMBEAU, MD,phD, Principal Investigator — Amiens Universitary Hospital
Locations (1):
- Amiens University Hospital, Amiens, France

REFERENCES:
- [Background] Pequignot A, Dhahria A, Mensah E, Verhaeghe P, Badaoui R, Sabbagh C, Regimbeau JM. Stapling and Section of the Nasogastric Tube during Sleeve Gastrectomy: How to Prevent and Recover? Case Rep Gastroenterol. 2011;5(2):350-4. doi: 10.1159/000329706. Epub 2011 Jul 6. PMID 21769286
- [Background] Dhahri A, Verhaeghe P, Hajji H, Fuks D, Badaoui R, Deguines JB, Regimbeau JM. Sleeve gastrectomy: technique and results. J Visc Surg. 2010 Oct;147(5 Suppl):e39-46. doi: 10.1016/j.jviscsurg.2010.08.016. No abstract available. PMID 20971049
- [Background] Sabbagh C, Verhaeghe P, Dhahri A, Brehant O, Fuks D, Badaoui R, Regimbeau JM. Two-year results on morbidity, weight loss and quality of life of sleeve gastrectomy as first procedure, sleeve gastrectomy after failure of gastric banding and gastric banding. Obes Surg. 2010 Jun;20(6):679-84. doi: 10.1007/s11695-009-0007-4. Epub 2009 Nov 10. PMID 19902316
- [Background] Fuks D, Verhaeghe P, Brehant O, Sabbagh C, Dumont F, Riboulot M, Delcenserie R, Regimbeau JM. Results of laparoscopic sleeve gastrectomy: a prospective study in 135 patients with morbid obesity. Surgery. 2009 Jan;145(1):106-13. doi: 10.1016/j.surg.2008.07.013. Epub 2008 Sep 30. PMID 19081482
- [Background] Fuks D, Dumont F, Berna P, Verhaeghe P, Sinna R, Sabbagh C, Demuynck F, Yzet T, Delcenserie R, Bartoli E, Regimbeau JM. Case report-complex management of a postoperative bronchogastric fistula after laparoscopic sleeve gastrectomy. Obes Surg. 2009 Feb;19(2):261-264. doi: 10.1007/s11695-008-9643-3. Epub 2008 Aug 12. PMID 18696169
- [Result] Deguines JB, Verhaeghe P, Yzet T, Robert B, Cosse C, Regimbeau JM. Is the residual gastric volume after laparoscopic sleeve gastrectomy an objective criterion for adapting the treatment strategy after failure? Surg Obes Relat Dis. 2013 Sep-Oct;9(5):660-6. doi: 10.1016/j.soard.2012.11.010. Epub 2013 Jan 17. PMID 23452922